CLINICAL TRIAL: NCT01800695
Title: A Phase 1 Study Evaluating the Safety and Pharmacokinetics of ABT-414 for Subjects With Glioblastoma Multiforme
Brief Title: Evaluating the Safety and Pharmacokinetics of ABT-414 for Subjects With Glioblastoma Multiforme
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M12-356; 2012-003884-23 (EudraCT Number)
Record Dates: First submitted 2013-02-05; First posted 2013-02-28 (Estimated); Last update posted 2017-11-21 (Actual); Status verified 2017-07

CONDITIONS: Glioblastoma Multiforme
Keywords: GBM
MeSH Terms: conditions — Glioblastoma | interventions — ABT-414; depatuxizumab mafodotin; Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Arm A (Experimental): ABT-414 in combination with radiation and temozolomide
  Interventions: Drug: ABT-414; Drug: Temozolomide; Radiation: Whole Brain Radiation
- Arm B (Experimental): ABT-414 in combination with temozolomide
  Interventions: Drug: ABT-414; Drug: Temozolomide
- Arm C (Experimental): ABT-414 monotherapy
  Interventions: Drug: ABT-414

INTERVENTIONS:
Drug: ABT-414 — ABT-414 will be administered by intravenous infusion
  Other Names: Depatuxizumab Mafodotin
Drug: Temozolomide — Temozolomide will be administered per label and local prescribing regulations.
  Arms: Arm A; Arm B
Radiation: Whole Brain Radiation — Whole Brain radiation will be administered in 30 fractions.
  Arms: Arm A

SUMMARY:
This study is evaluating the safety and pharmacokinetics of ABT-414 in subjects with glioblastoma multiforme.

ELIGIBILITY:
Inclusion Criteria:

1. Glioblastoma Multiforme (GBM)
2. 70 or above on Karnofsky Performance Status
3. Adequate bone marrow function
4. Recurrent GBM per RANO criteria
5. Subjects must have confirmed EGFR amplification by central lab

Exclusion Criteria:

1. For Subjects with recurrent GBM in Arm B, subject has received prior treatment with bevacizumab, nitrosourea, or has secondary GBM
2. For Subjects with recurrent GBM in Arm C, subject has received prior treatment with bevacizumab, or has secondary GBM
3. Allergies to temozolomide, dacarbazine, IgG containing agents
4. Anti-cancer treatment 28 days prior to study Day 1, except in Arm B expanded cohort temozolomide therapy is allowed
5. Subjects that have had more than one disease recurrence

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2013-04-02 (Actual); Primary Completion 2017-06-19 (Actual); Study Completion 2017-06-19 (Actual)

PRIMARY OUTCOMES:
Number and percentage of participants with adverse events | Every week for an expected average of 34 weeks
  Measurement by clinical lab results, vital signs, physical exam, and electrocardiogram (ECG)
Maximum concentration of ABT-414 | Multiple time points in Cycles 1, 2, and 3 (4 weeks each) and Day 1 of remaining cycles until end of treatment, an expected average of 34 weeks
  Measurement of the maximum concentration of ABT- 414 in the blood
Number of Dose Limiting Toxicities | Every week for an expected average of 34 weeks
  Measurement by clinical lab results, vital signs, physical exam, and electrocardiogram (ECG)
Minimum Concentration of ABT-414 | Multiple time points in Cycles 1, 2, and 3 (4 weeks each) and Day 1 of remaining cycles until end of treatment, an expected average of 34 weeks
  Measurement of the minimum concentration of ABT-414 in the blood
Half-life of ABT-414 | Multiple time points in Cycles 1, 2, and 3 (4 weeks each) and Day 1 of remaining cycles until end of treatment, an expected average of 34 weeks
  Measurement of the clearance of ABT-414

SECONDARY OUTCOMES:
Biomarker EGFR expression | At screening and post-study
  Assessment of tumor biomarkers that may correlate with efficacy.
Progression Free Survival | Multiple time points in each cycle, throughout study, and survival information monthly until 1 year after last visit, or the participant becomes lost to follow up, or study termination.
  Progression Free Survival per RANO criteria is the length of time during and after the treatment of a disease, that the participant lives with the disease but does not get worse.
Overall Survival | Multiple time points in each cycle, throughout study, and survival information monthly until 1 year after last visit, or participant becomes lost to follow up, or study termination
  The overall response rate will be evaluated every 8 weeks at each assessment of disease according to RANO criteria, up to 28 months

CONTACTS AND LOCATIONS:
Overall Officials: Earle Bain, MD, Study Director — AbbVie

REFERENCES:
- [Derived] Lassman AB, Roberts-Rapp L, Sokolova I, Song M, Pestova E, Kular R, Mullen C, Zha Z, Lu X, Gomez E, Bhathena A, Maag D, Kumthekar P, Gan HK, Scott AM, Guseva M, Holen KD, Ansell PJ, van den Bent MJ. Comparison of Biomarker Assays for EGFR: Implications for Precision Medicine in Patients with Glioblastoma. Clin Cancer Res. 2019 Jun 1;25(11):3259-3265. doi: 10.1158/1078-0432.CCR-18-3034. Epub 2019 Feb 22. PMID 30796037
- [Derived] Lassman AB, van den Bent MJ, Gan HK, Reardon DA, Kumthekar P, Butowski N, Lwin Z, Mikkelsen T, Nabors LB, Papadopoulos KP, Penas-Prado M, Simes J, Wheeler H, Walbert T, Scott AM, Gomez E, Lee HJ, Roberts-Rapp L, Xiong H, Ansell PJ, Bain E, Holen KD, Maag D, Merrell R. Safety and efficacy of depatuxizumab mafodotin + temozolomide in patients with EGFR-amplified, recurrent glioblastoma: results from an international phase I multicenter trial. Neuro Oncol. 2019 Jan 1;21(1):106-114. doi: 10.1093/neuonc/noy091. PMID 29982805
- [Derived] Goss GD, Vokes EE, Gordon MS, Gandhi L, Papadopoulos KP, Rasco DW, Fischer JS, Chu KL, Ames WW, Mittapalli RK, Lee HJ, Zeng J, Roberts-Rapp LA, Loberg LI, Ansell PJ, Reilly EB, Ocampo CJ, Holen KD, Tolcher AW. Efficacy and safety results of depatuxizumab mafodotin (ABT-414) in patients with advanced solid tumors likely to overexpress epidermal growth factor receptor. Cancer. 2018 May 15;124(10):2174-2183. doi: 10.1002/cncr.31304. Epub 2018 Mar 13. PMID 29533458